CLINICAL TRIAL: NCT04959201
Title: Combination of NMDA-enhancing and Antioxidant Treatments for Schizophrenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH108-REC1-177
Record Dates: First submitted 2021-06-10; First posted 2021-07-13 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; NMDA; Oxidative stress
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMDAE plus Antioxidant agent (AO) (Experimental): An NMDA enhancer plus a drug with antioxidant property
  Interventions: Drug: NMDAE plus AO
- NMDAE plus Placebo (Placebo Comparator): An NMDA enhancer plus Placebo
  Interventions: Drug: NMDAE plus Placebo Cap

INTERVENTIONS:
Drug: NMDAE plus AO — Use of an NMDA enhancer plus a drug with antioxidant property for the treatment of schizophrenia.
  Arms: NMDAE plus Antioxidant agent (AO)
Drug: NMDAE plus Placebo Cap — Use of an NMDA enhancer plus placebo as a comparator.
  Arms: NMDAE plus Placebo

SUMMARY:
Previous studies found that some NMDA-enhancing agents were able to improve clinical symptoms of patients with schizophrenia. In addition, several drugs with antioxidant properties have been tested in clinical trials for the treatment of schizophrenia too. Whether combined treatment of an NMDA-enhancing agent and a drug with antioxidant property can be better than an NMDA-enhancing agent alone deserves study.

DETAILED DESCRIPTION:
Several lines of evidence suggest that both NMDA and oxidative stress hypotheses have been implicated in schizophrenia. Previous studies found that some NMDA-enhancing agents were able to augment efficacy of antipsychotics in the treatment of schizophrenia. In addition, several drugs with antioxidant properties have been tested in clinical trials for the treatment of schizophrenia too. Whether a drug with antioxidant property can strengthen the efficacy of an NMDA-enhancer (NMDAE) in the treatment of schizophrenia remains unknown. Therefore, this study aims to compare NMDAE plus a drug with antioxidant property and NMDAE plus placebo in the treatment of schizophrenia. The subjects are the schizophrenia patients who remain symptomatic while having been stabilized with antipsychotic treatment. They keep their original treatment and are randomly, double-blindly assigned into two treatment groups for 12 weeks: (1) NMDAE plus Antioxidant agent (AO), or (2) NMDAE plus placebo. Clinical performances and side effects are measured at weeks 0, 2, 4, 6, 9, and 12. Cognitive functions are assessed at baseline and at endpoint of treatment by a battery of tests. The efficacies of NMDAE plus AO and NMDAE plus placebo will be compared.

Chi-square (or Fisher's exact test) will be used to compare differences of categorical variables and t-test (or Mann-Whitney test if the distribution is not normal) for continuous variables between treatment groups. Mean changes from baseline in repeated-measure assessments will be assessed using the generalized estimating equation (GEE). All p values for clinical measures will be based on two-tailed tests with a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Have a DSM-5 (American Psychiatric Association) diagnosis of schizophrenia
* Remain symptomatic but without clinically significant fluctuation, while their antipsychotic doses are unchanged for at least 3 months and will be maintained during the period of the 12-week trial
* PANSS total score ≥ 60
* Agree to participate in the study and provide informed consent

Exclusion Criteria:

* DSM-5 diagnosis of intellectual disability or substance (including alcohol) use disorder
* History of epilepsy, head trauma, stroke, or serious medical or central nervous system diseases (other than schizophrenia) which may interfere with the study
* Clinically significant laboratory screening tests (including blood routine, biochemical tests)
* Pregnancy or lactation
* Inability to follow protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change of Positive and Negative Syndrome Scale (PANSS) | week 0, 2, 4, 6, 9, 12
  Assessment of overall symptoms. Minimum value: 30, maximum value:210, the higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change of scales for the Assessment of Negative Symptoms (SANS) total score | week 0, 2, 4, 6, 9, 12
  Assessment of negative symptoms. Minimum value: 0, maximum value:100, the higher scores mean a worse outcome.
Positive subscale of PANSS | week 0, 2, 4, 6, 9, 12
  Assessment of positive symptoms. Minimum value: 7, maximum value:49, the higher scores mean a worse outcome.
Negative subscale of PANSS | week 0, 2, 4, 6, 9, 12
  Assessment of negative symptoms. Minimum value: 7, maximum value:49, the higher scores mean a worse outcome.
General Psychopathology subscale of PANSS | week 0, 2, 4, 6, 9, 12
  Assessment of general psychopathology. Minimum value: 16, maximum value:112, the higher scores mean a worse outcome.
Clinical Global Impression | week 0, 2, 4, 6, 9, 12
  Assessment of general impression. Minimum value: 1, maximum value:7, the higher scores mean a worse outcome.
Global Assessment of Functioning | week 0, 2, 4, 6, 9, 12
  Assessment of social, occupational, and psychological function. Minimum value: 1, maximum value:100, the higher scores mean better function.
Hamilton Rating Scale for Depression | week 0, 2, 4, 6, 9, 12
  Assessment of depressive symptoms. Minimum value: 0, maximum value:52, the higher scores mean a worse outcome
Quality of Life Scale | week 0, 2, 4, 6, 9, 12
  Assessment of life quality. Minimum value: 0, maximum value:126, the higher scores mean a better outcome.
Cognitive function | Week 0, 12
  Ten tests for assessment of 7 cognitive domains:
  1. speed of processing (assessed by Category Fluency, Trail Marking A, WAIS-III Digit Symbol-Coding)
  2. sustained attention (Continuous Performance Test)
  3. working memory: verbal (digit span) and nonverbal (spatial span)
  4. verbal learning and memory (WMS-III, word listing)
  5. visual learning and memory (WMS-III, visual reproduction)
  6. reasoning and problem solving (WISC-III, Maze)
  7. social cognition (MSCEIT Version 2)
  All tests have no unit. Firstly, for the domain (a. and c.) with more than one test, a composite T score will be calculated by standardizing the average of each T score (with a mean of 50 and a SD of 10 for making every test comparative). Secondly, a global composite score (for all seven domains) and a neurocognitive composite score (for the first 6 domains, a-f) will be also calculated by standardizing the average of the T score of each domain (Lane HY et al, JAMA Psychiatry. 2013).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, China Medical University Hospital, Taichung, Taiwan